CLINICAL TRIAL: NCT02772276
Title: A Pilot Safety and Pharmacokinetic Study of MB-102 Versus Iohexol and the Use of the Non-invasive Optical Renal Function Monitor (ORFM) Device in Subjects With Normal and Impaired Renal Function and a Range of Skin Color Types
Brief Title: Pharmacokinetics of MB-102 and Use of the Non-invasive Optical Renal Function Monitor (ORFM) Device in Subjects With Normal and Impaired Renal Function and a Range of Skin Color Types
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediBeacon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ORFM-2
Record Dates: First submitted 2016-05-10; First posted 2016-05-13 (Estimated); Results first posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Acute Kidney Injury
Keywords: Glomerular Filtration Rate
MeSH Terms: conditions — Acute Kidney Injury | interventions — relmapirazin; Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (13):
- Normal-CKD Stage 2/QuantumLeap (Experimental): MB-102 and iohexol administered to participants with normal to chronic kidney disease (CKD) Stage 2 renal function, and fluorescence measured by the QuantumLeap ORFM device. Approximately half of the participants were to be enrolled with Fitzpatrick Scale Type I, II or III, and half with Type IV, V and VI skin color type. In order to determine the optimal dose of MB-102, participants may have received different doses.
  Interventions: Drug: MB-102-- single dose of 4 µmol/kg; Drug: Iohexol; Device: QuantumLeap
- CKD Stage 3-4/QuantumLeap (Experimental): MB-102 and iohexol administered to participants with impaired renal function (chronic kidney disease (CKD) Stage 3-4), and fluorescence measured by the QuantumLeap ORFM device. Approximately half of the participants were to be enrolled with Fitzpatrick Scale Type I, II or III, and half with Type IV, V and VI skin color type. In order to determine the optimal dose of MB-102, participants may have received different doses.
  Interventions: Drug: MB-102-- single dose of 4 µmol/kg; Drug: Iohexol; Device: QuantumLeap
- Normal-CKD Stage 2/Radiance (Experimental): MB-102 and iohexol administered to participants with normal to chronic kidney disease (CKD) Stage 2 renal function, and fluorescence measured by the Radiance ORFM device. Approximately half of the participants were to be enrolled with Fitzpatrick Scale Type I, II or III, and half with Type IV, V and VI skin color type.
  Interventions: Drug: MB-102-- single dose of 4 µmol/kg; Drug: Iohexol; Device: Radiance
- CKD Stage 3-5/Radiance (Experimental): MB-102 and iohexol administered to participants with impaired renal function (chronic kidney disease (CKD) Stage 3-5), and fluorescence measured by the Radiance ORFM device. Approximately half of the participants were to be enrolled with Fitzpatrick Scale Type I, II or III, and half with Type IV, V and VI skin color type.
  Interventions: Drug: MB-102-- single dose of 4 µmol/kg; Drug: Iohexol; Device: Radiance
- Normal-CKD Stage 2/Brilliance algorithm optimization (Experimental): MB-102 administered to participants with normal to chronic kidney disease (CKD) Stage 2 renal function, and fluorescence measured by the Brilliance ORFM device. Algorithm optimization of the Brilliance sensor was conducted. Approximately half of the participants were to be enrolled with Fitzpatrick Scale Type I, II or III, and half with Type IV, V and VI skin color type.
  Interventions: Drug: MB-102-- single dose of 4 µmol/kg; Device: Brilliance (1 or 2 sensors)
- CKD Stage 3-5/Brilliance algorithm optimization (Experimental): MB-102 administered to participants with impaired renal function (chronic kidney disease (CKD) Stage 3-5), and fluorescence measured by the Brilliance ORFM device. Algorithm optimization of the Brilliance sensor was conducted. Approximately half of the participants were to be enrolled with Fitzpatrick Scale Type I, II or III, and half with Type IV, V and VI skin color type.
  Interventions: Drug: MB-102-- single dose of 4 µmol/kg; Device: Brilliance (1 or 2 sensors)
- Normal-CKD Stage 2/Brilliance sensor optimization (Experimental): MB-102 administered to participants with normal to chronic kidney disease (CKD) Stage 2 renal function, and fluorescence measured by the Brilliance ORFM device. Sensor optimization of the Brilliance device was conducted. Approximately half of the participants were to be enrolled with Fitzpatrick Scale Type I, II or III, and half with Type IV, V and VI skin color type.
  Interventions: Drug: MB-102-- single dose of 4 µmol/kg; Device: Brilliance (1 or 2 sensors)
- Normal-CKD Stage 2/Brilliance sensor validation (Experimental): MB-102 administered to participants with normal to chronic kidney disease (CKD) Stage 2 renal function, and fluorescence measured by the Brilliance ORFM device. Validation of the Brilliance sensor was conducted. Approximately half of the participants were to be enrolled with Fitzpatrick Scale Type I, II or III, and half with Type IV, V and VI skin color type.
  Interventions: Drug: MB-102-- single dose of 4 µmol/kg; Device: Brilliance (1 or 2 sensors)
- CKD Stage 3-5/Brilliance sensor validation (Experimental): MB-102 administered to participants with impaired renal function (chronic kidney disease (CKD) Stage 3-5), and fluorescence measured by the Brilliance ORFM device. Validation of the Brilliance sensor was conducted. Approximately half of the participants were to be enrolled with Fitzpatrick Scale Type I, II or III, and half with Type IV, V and VI skin color type.
  Interventions: Drug: MB-102-- single dose of 130 mg; Device: Brilliance (1 or 2 sensors)
- Normal-CKD Stage 2/Brilliance (1-2 sensors) (Experimental): MB-102 administered to participants with normal to chronic kidney disease (CKD) Stage 2 renal function, and fluorescence measured by the Brilliance ORFM device (1-2 sensors). The optimized algorithm and final device design of the Brilliance device was tested. Approximately half of the participants were to be enrolled with Fitzpatrick Scale Type I, II or III, and half with Type IV, V and VI skin color type. A subset of participants in this arm received two doses of MB-102, 12 hours apart.
  Interventions: Drug: MB-102-single dose of 130 mg or 2 doses of 130 mg 12 hours apart; Device: Brilliance (1 or 2 sensors)
- Normal-CKD Stage 2/Brilliance (1-2 sensors and Brilliance 2-part sensor) (Experimental): MB-102 administered to participants with normal to chronic kidney disease (CKD) Stage 2 renal function, and fluorescence measured by the Brilliance ORFM device (1-2 sensors and 2-part sensor). The optimized algorithm and final device design of the Brilliance device was tested. Approximately half of the participants were to be enrolled with Fitzpatrick Scale Type I, II or III, and half with Type IV, V and VI skin color type. A subset of participants in this arm received two doses of MB-102, 12 hours apart.
  Interventions: Drug: MB-102-single dose of 130 mg or 2 doses of 130 mg 12 hours apart; Device: Brilliance (1 or 2 sensors); Device: Brilliance (2-part sensor)
- Normal-CKD Stage 2/Brilliance (1-2 sensors and Brilliance 2-part sensor) and 2 doses MB-102 (Experimental): Two doses of MB-102 administered to participants 12 hours apart, with normal to chronic kidney disease (CKD) Stage 2 renal function, and fluorescence measured by the Brilliance ORFM device (1-2 sensors and 2-part sensor). The optimized algorithm and final device design of the Brilliance device was tested. Approximately half of the participants were to be enrolled with Fitzpatrick Scale Type I, II or III, and half with Type IV, V and VI skin color type.
  Interventions: Drug: MB-102-- two doses of 130 mg 24 hours apart; Device: Brilliance (1 or 2 sensors); Device: Brilliance (2-part sensor)
- CKD Stage 3-5/Brilliance 1-2 sensors (Experimental): MB-102 administered to participants with impaired renal function (chronic kidney disease (CKD) Stage 3-5), and fluorescence measured by the Brilliance ORFM device. The optimized algorithm and final device design of the Brilliance device was tested. Approximately half of the participants were to be enrolled with Fitzpatrick Scale Type I, II or III, and half with Type IV, V and VI skin color type.
  Interventions: Drug: MB-102-- single dose of 130 mg; Device: Brilliance (1 or 2 sensors)

INTERVENTIONS:
Drug: MB-102-- single dose of 4 µmol/kg — 4 µmol/kg administered by intravenous injection over 30 seconds, followed by a 10 mL normal saline flush administered intravenously over 30 seconds.
  Other Names: Relmapirazin
  Arms: CKD Stage 3-4/QuantumLeap; CKD Stage 3-5/Brilliance algorithm optimization; CKD Stage 3-5/Radiance; Normal-CKD Stage 2/Brilliance algorithm optimization; Normal-CKD Stage 2/Brilliance sensor optimization; Normal-CKD Stage 2/Brilliance sensor validation; Normal-CKD Stage 2/QuantumLeap; Normal-CKD Stage 2/Radiance
Drug: MB-102-- single dose of 130 mg — 130 mg administered by intravenous injection over 30 seconds, followed by a 10 mL normal saline flush administered intravenously over 30 seconds. A subset of participants will receive two doses of MB-102, 12 hours apart.
  Other Names: Relmapirazin
  Arms: CKD Stage 3-5/Brilliance 1-2 sensors; CKD Stage 3-5/Brilliance sensor validation
Drug: MB-102-single dose of 130 mg or 2 doses of 130 mg 12 hours apart — 130 mg administered by intravenous injection over 30 seconds, followed by a 10 mL normal saline flush administered intravenously over 30 seconds.
  Other Names: Relmapirazin
  Arms: Normal-CKD Stage 2/Brilliance (1-2 sensors and Brilliance 2-part sensor); Normal-CKD Stage 2/Brilliance (1-2 sensors)
Drug: MB-102-- two doses of 130 mg 24 hours apart — 4 µmol/kg administered by intravenous injection over 30 seconds, followed by a 10 mL normal saline flush administered intravenously over 30 seconds. A subset of participants will receive two doses of MB-102, 12 hours apart.
  Other Names: Relmapirazin
  Arms: Normal-CKD Stage 2/Brilliance (1-2 sensors and Brilliance 2-part sensor) and 2 doses MB-102
Drug: Iohexol — 5 mL of a 647 mg/mL solution administered by intravenous injection over 30 seconds, followed by a 10 mL normal saline flush administered intravenously over 30 seconds
  Other Names: Omnipaque 300
  Arms: CKD Stage 3-4/QuantumLeap; CKD Stage 3-5/Radiance; Normal-CKD Stage 2/QuantumLeap; Normal-CKD Stage 2/Radiance
Device: QuantumLeap — Optical Renal Function Monitor (ORFM)
  Arms: CKD Stage 3-4/QuantumLeap; Normal-CKD Stage 2/QuantumLeap
Device: Radiance — Optical Renal Function Monitor (ORFM)
  Arms: CKD Stage 3-5/Radiance; Normal-CKD Stage 2/Radiance
Device: Brilliance (1 or 2 sensors) — Optical Renal Function Monitor (ORFM)
  Arms: CKD Stage 3-5/Brilliance 1-2 sensors; CKD Stage 3-5/Brilliance algorithm optimization; CKD Stage 3-5/Brilliance sensor validation; Normal-CKD Stage 2/Brilliance (1-2 sensors and Brilliance 2-part sensor); Normal-CKD Stage 2/Brilliance (1-2 sensors and Brilliance 2-part sensor) and 2 doses MB-102; Normal-CKD Stage 2/Brilliance (1-2 sensors); Normal-CKD Stage 2/Brilliance algorithm optimization; Normal-CKD Stage 2/Brilliance sensor optimization; Normal-CKD Stage 2/Brilliance sensor validation
Device: Brilliance (2-part sensor) — Optical Renal Function Monitor (ORFM)
  Arms: Normal-CKD Stage 2/Brilliance (1-2 sensors and Brilliance 2-part sensor); Normal-CKD Stage 2/Brilliance (1-2 sensors and Brilliance 2-part sensor) and 2 doses MB-102

SUMMARY:
This study was a pilot, safety, and pharmacokinetic study of MB-102 versus iohexol and the use of the non-invasive optical renal function monitor (ORFM) device in normal and compromised renal function participants with different skin color types.

DETAILED DESCRIPTION:
The objectives of this study were to evaluate the safety and tolerability of single and multiple doses of MB-102 in participants with normal and impaired kidney function; to determine plasma pharmacokinetics of MB-102 compared to the pharmacokinetics of iohexol in participants with normal and impaired kidney function; to demonstrate that MB-102-transdermal-fluorescence-measured glomerular filtration rate (GFR) using the optical renal function monitor (ORFM) Brilliance device is aligned with MB-102 plasma GFR; to evaluate the safety and effectiveness of the ORFM investigational medical device prototypes QuantumLeap, Radiance, and Brilliance for the non-invasive transdermal fluorescent detection of MB-102 in participants with a range of skin color types; and to determine the optimal dose of MB-102 for non-invasive measurement.

ELIGIBILITY:
INCLUSION CRITERIA

Main Criteria for Inclusion (Quantum Leap and Radiance device)

* Age > 22 years - male or female

  * Eligible female non-pregnant participants who are either not of childbearing potential or willing to use adequate contraception during the trial
  * Males must be willing to practice abstinence or utilize adequate contraception from dosing day to at least 7 days post dose
* Participants willing to comply with study requirements
* Participants who have signed an informed consent form
* Normal or non-clinically significant screening and baseline 12-lead electrocardiogram (ECG) in the opinion of the principal investigator (PI)
* Adequate venous access sufficient to allow blood sampling per protocol requirements

Main Criteria for Inclusion (Brilliance device)

* Age > 18 years - male or female

  * Eligible female non-pregnant participants who are either not of childbearing potential or willing to use adequate contraception during the trial
  * Males must be willing to practice abstinence or utilize adequate contraception from dosing day to at least 7 days post dose
* Participants willing to comply with study requirements
* Participants who have signed an informed consent form
* Normal or non-clinically significant screening and baseline 12-lead ECG in the opinion of the PI
* Adequate venous access sufficient to allow blood sampling per protocol requirements

Normal-CKD Stage 2/QuantumLeap; Normal-CKD Stage 2/Radiance; Normal-CKD Stage 2/Brilliance algorithm optimization; Normal-CKD Stage 2/Brilliance sensor optimization; Normal-CKD Stage 2/Brilliance sensor optimization; and Normal-CKD Stage 2/Brilliance (1-2 sensors)

* Are healthy as determined by medical history, with no clinically significant findings on screening and baseline physical exams, vital signs and clinical laboratory panels or conditions that could adversely impact the participant's participation or safety, conduct of the study or interfere with study assessments
* Have estimated glomerular filtration rate (eGFR (Chronic kidney disease - epidemiology collaboration [CKD-EPI] equation) of ≥60 ml/min/1.73m^2 (normal to Stage 2 CKD) at the time of screening
* Approximately half of the participants enrolled in each cohort to have Fitzpatrick Scale Type I, II or III skin color type
* Approximately half of the participants enrolled in each cohort to have Fitzpatrick Type IV, V or VI skin color type.

CKD Stage 3-4/QuantumLeap

* Possess stable renal function in the opinion of the PI
* Have eGFR (CKD-EPI equation) of 15 - 59 mL/min/1.73m^2 at the time of screening
* Stable use of immunosuppressant medications (when applicable)

  * 15 participants per cohort to have Fitzpatrick Type I, II or III skin color type
  * 15 participants per cohort to have Fitzpatrick Type IV, V or VI skin color type

CKD Stage 3-5/Radiance; CKD Stage 3-5/Brilliance algorithm optimization; CKD Stage 3-5/Brilliance sensor validation; and CKD Stage 3-5/Brilliance 1-2 sensors

* Possess stable renal function as defined as the most recent historical (within 3 months) eGFR and screening eGFR differing by ≤20%.
* Have eGFR (CKD-EPI equation) of <59 mL/min/1.73m^2 based on a historical value collected within 3 months or from the screening serum creatinine
* Stable use of immunosuppressant medications (when applicable) defined as no changes in the last 30 days or expected through the follow up visits, and a prednisone dose of <20 mg/day (or another steroid's equivalent dose)
* Approximately half of the participants in each cohort to have Fitzpatrick Type I, II or III skin color type
* Approximately half of the participants in each cohort to have Fitzpatrick Type IV, V or VI skin color type

EXCLUSION CRITERIA

Main Criteria for Exclusion (QuantumLeap device)

* Women who are pregnant, lactating or planning to become pregnant during the study, or women who are of childbearing potential unwilling to use a barrier method of birth control
* Intolerant to venipuncture
* Recent donation or loss of blood or plasma: 100 mL to 499 mL within 30 days prior to the initial dose of the study medication; or more than 499 mL within 56 days prior to the initial dose of study medication
* Participation in another interventional trial within 30 days of screening or concurrently enrolled in any other medical research study which could impact the results of the study
* History of drug or alcohol abuse within the past year
* History of allergy or hypersensitivity to MB-102 or iohexol, or other related (iodinated contrast media) products, or any of the inactive ingredients
* History of skin sensitivity to adhesives (e.g. Band-Aids, surgical tape)
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the PI, could contraindicate the subject's participation in this study
* Participants who have allergies to 2 or more classes of drugs. (Intolerance to a drug is not considered a drug allergy)
* Stable use (no changes within 30 days) of prescription or over the counter (OTC) medications
* Non-steroidal anti-inflammatory drug (NSAID) use within 2 days of dosing day
* History of coagulation disorders or bleeding disorders that in the judgement of the investigator places the subject at undue risks for study related procedures
* Are homozygous for sickle cell disease
* Have a known thyroid disorder
* Have pheochromocytoma
* Currently on Coumadin (warfarin) who have an International normalized ratio (INR) >4 at Screening
* Current history of AIDS or HIV
* Hepatitis B antigen positive, or C antibody positive
* Site personnel immediately associated with the study or their immediate family members
* Any characteristics which, in the opinion of the investigator, makes the participant a poor candidate for participation in the clinical trial
* Prior enrollment and dosing in this Pilot 2 study
* Significant scaring, tattoos or alterations in pigmentation on the sternum that would alter sensor readings versus other areas of the skin

Additional Exclusion: Normal-CKD Stage 2/QuantumLeap

• History of significant cardiovascular disease, heart failure, myocardial infarction in the past 3 months, pulmonary, hematologic, endocrine, hepatobiliary, nephrologic, immunologic, dermatologic, neurologic (including any history of stroke and/or seizure disorder), psychological, musculoskeletal disease, diagnosis of cancer with the past 2 years or deemed clinically significant or unstable by the Principal Investigator; Note: history of gallstones or kidney stones are not excluded so long as the condition is not acute within 30 days of dosing.

Additional Exclusion: CKD Stage 3-4/QuantumLeap

* Stage 5 CKD at the time of screening
* Recent (within 3 months) significant medical condition or surgical procedure including myocardial infarction, laparoscopic procedures, or other medical inventions
* Doses of prednisone greater than 10 mg/day within the last 90 days

Main Criteria for Exclusion: (Radiance device)

* Women who are pregnant, lactating or planning to become pregnant during the study, or women who are of childbearing potential unwilling to use a barrier method of birth control

  o Males must be willing to practice abstinence or utilize adequate contraception from dosing day to at least 7 days post dose
* Unable to have venous access placed in both arms
* Recent donation or loss of blood or plasma: 100 mL to 499 mL within 30 days prior to the initial dose of the study medication; or more than 499 mL within 56 days prior to the initial dose of study medication
* Participation in another interventional trial within 30 days of dosing or concurrently enrolled in any other medical research study which could impact the results of the study
* History of drug or alcohol abuse within the past year
* History of skin sensitivity to adhesives (e.g. Band-Aids, surgical tape)
* History of severe allergic hypersensitivity reactions (unacceptable adverse events) or anaphylactoid reaction to any allergen including drugs, MB-102 and iohexol or other related (iodinated contrast media) products (intolerance to a drug is not considered a drug allergy)
* NSAID use within 2 days of dosing day
* History of coagulation disorders or bleeding disorders that in the judgement of the investigator places the subject at undue risks for study related procedures
* Are homozygous for sickle cell disease
* Have hyperthyroidism or current thyroid cancer
* Have pheochromocytoma
* Currently on Coumadin (warfarin) who have an INR >4 at Screening
* Current history of AIDS or HIV
* Current evidence of an active Hepatitis B or C infection. If the participant is Hepatitis C antibody positive, but the hepatitis C RNA is below the level of detection, they are considered immune and may be eligible for enrollment.
* Site personnel immediately associated with the study or their immediate family members
* Any characteristics which, in the opinion of the investigator, makes the subject a poor candidate for participation in the clinical trial
* Prior exposure to MB-102
* Significant scaring, tattoos or alterations in pigmentation on the sternum that would alter sensor readings versus other areas of the skin

Main Criteria for Exclusion: (Brilliance device)

* Women who are pregnant, lactating or planning to become pregnant during the study, or women who are of childbearing potential unwilling to use a barrier method of birth control

  o Males must be unwilling to practice abstinence or utilize adequate contraception from dosing day to at least 7 days post dose
* Unable to have venous access
* Recent donation or loss of blood or plasma: 100 mL to 499 mL within 30 days prior to the initial dose of the study medication; or more than 499 mL within 56 days prior to the initial dose of study medication
* Participation in another interventional trial within 30 days of dosing or concurrently enrolled in any other medical research study which could impact the results of the study
* History of drug or alcohol abuse within the past year
* History of skin sensitivity to adhesives (e.g. Band-Aids, surgical tape)
* History of severe allergic hypersensitivity reactions (unacceptable adverse events) or anaphylactoid reaction to any allergen including drugs, or MB-102 (intolerance to a drug is not considered a drug allergy)
* NSAID use within 2 days of dosing day
* History of coagulation disorders or bleeding disorders that in the judgement of the investigator places the subject at undue risks for study related procedures
* Currently on Coumadin (warfarin) who have an INR >4 at Screening
* Current history of AIDS or HIV
* Current evidence of an active Hepatitis B or C infection. If the participant is Hepatitis C antibody positive, but the hepatitis C RNA is below the level of detection, they are considered immune and may be eligible for enrollment.
* Site personnel immediately associated with the study or their immediate family members
* Any characteristics which, in the opinion of the investigator, makes the participant a poor candidate for participation in the clinical trial
* Significant scaring, tattoos or alterations in pigmentation on the sternum that would alter sensor readings versus other areas of the skin

Additional Exclusion: Normal-CKD Stage 2/Radiance; Normal-CKD Stage 2/Brilliance algorithm optimization; Normal-CKD Stage 2/Brilliance sensor optimization; Normal-CKD Stage 2/Brilliance sensor validation; and Normal-CKD Stage 2/Brilliance (1-2 sensors)

* History of significant cardiovascular disease, heart failure, myocardial infarction in the past 3 months, or NYHA class III or IV HF
* Any other serious or uncontrolled medical disorder, active infection, physical exam finding, laboratory finding, or psychiatric condition that in the opinion of the investigator would limit the participant's ability to complete study requirements or may put the subject at increased risk or compromise interpretability of study results. Note: a history of gallstones or kidney stones are not excluded so long as the condition is not acute within 30 days of dosing.

Additional Exclusion: CKD Stage 3-5/Radiance; CKD Stage 3-5/Brilliance algorithm optimization; CKD Stage 3-5/Brilliance sensor validation; and CKD Stage 3-5/Brilliance 1-2 sensors

* Recent (within 3 months) significant medical condition or surgical procedure including myocardial infarction, thoracic laparoscopic procedures, or other significant medical inventions
* Received >20 mg/day of prednisone or an equivalent dose of glucocorticoid for more than 7 days in the last 90 days prior to dosing day for an acute or chronic disorder
* Currently receiving dialysis
* Currently anuric

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Dorshow, PhD, Study Director — MediBeacon, Inc.
Locations (3):
- United States (3):
  - Riverside Clinical Research, Edgewater, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dorshow RB, Debreczeny MP, Goldstein SL. GFR Measurement Using Transdermal Detection Methodology. J Am Soc Nephrol. 2025 Feb 7;36(8):1592-1602. doi: 10.1681/ASN.0000000639. PMID 39918882

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Safety Analysis Set: all participants who signed the informed consent form and received study drug
Period: Overall Study
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance | Normal-CKD Stage 2/Brilliance Algorithm Optimization | CKD Stage 3-5/Brilliance Algorithm Optimization | Normal-CKD Stage 2/Brilliance Sensor Optimization | Normal-CKD Stage 2/Brilliance Sensor Validation | CKD Stage 3-5/Brilliance Sensor Validation | Normal-CKD Stage 2/Brilliance (1-2 Sensors) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) and 2 Doses MB-102 | CKD Stage 3-5/Brilliance 1-2 Sensors
Started | 31 | 29 | 20 | 40 | 9 | 7 | 18 | 30 | 18 | 12 | 4 | 4 | 12
Completed | 31 | 29 | 20 | 40 | 9 | 7 | 17 | 29 | 18 | 12 | 4 | 4 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who signed the informed consent form and received study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance | Normal-CKD Stage 2/Brilliance Algorithm Optimization | CKD Stage 3-5/Brilliance Algorithm Optimization | Normal-CKD Stage 2/Brilliance Sensor Optimization | Normal-CKD Stage 2/Brilliance Sensor Validation | CKD Stage 3-5/Brilliance Sensor Validation | Normal-CKD Stage 2/Brilliance (1-2 Sensors) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) and 2 Doses MB-102 | CKD Stage 3-5/Brilliance 1-2 Sensors | Total
Number analyzed (Participants) | 31 | 29 | 20 | 40 | 9 | 7 | 18 | 30 | 18 | 12 | 4 | 4 | 12 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (11.78) | 58.2 (11.76) | 54.7 (13.57) | 61.1 (12.93) | 46.9 (13.40) | 66.9 (6.67) | 41.6 (15.42) | 39.1 (15.38) | 70.9 (8.09) | 47.9 (17.70) | 52.3 (14.27) | 42.5 (13.72) | 70.3 (9.46) | 53 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 10 | 21 | 2 | 6 | 8 | 16 | 6 | 6 | 1 | 2 | 4 | 115
  Male | 12 | 15 | 10 | 19 | 7 | 1 | 10 | 14 | 12 | 6 | 3 | 2 | 8 | 119
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 15 | 11 | 7 | 15 | 4 | 2 | 7 | 11 | 1 | 6 | 2 | 2 | 4 | 87
  White | 15 | 18 | 11 | 25 | 5 | 5 | 11 | 19 | 17 | 6 | 2 | 2 | 8 | 144
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 29 | 20 | 40 | 9 | 7 | 18 | 30 | 18 | 12 | 4 | 4 | 12 | 234

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: An adverse event is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, temporally associated with the use of a medicinal product, whether or not related to the investigational medical device or drug.
Time Frame: From the time of dosing through the follow-up visit, up to 10 days
Population: Safety Analysis Set: all participants who signed the informed consent form and received study drug
Measure: Count of Participants; unit: Participants
Groups:
- Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor): MB-102 administered to participants with normal to chronic kidney disease (CKD) Stage 2 renal function,and fluorescence measured by the Brilliance ORFM device (1-2 sensors and 2-part sensor). The optimized algorithm and final device design of the Brilliance device was tested. Approximately half of the participants were to be enrolled with Fitzpatrick Scale Type I, II or III, and half with Type IV, V and VI skin color type. A subset of participants in this arm received two doses of MB-102, 12 hours apart.
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance | Normal-CKD Stage 2/Brilliance Algorithm Optimization | CKD Stage 3-5/Brilliance Algorithm Optimization | Normal-CKD Stage 2/Brilliance Sensor Optimization | Normal-CKD Stage 2/Brilliance Sensor Validation | CKD Stage 3-5/Brilliance Sensor Validation | Normal-CKD Stage 2/Brilliance (1-2 Sensors) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) and 2 Doses MB-102 | CKD Stage 3-5/Brilliance 1-2 Sensors
Number analyzed (Participants) | 31 | 29 | 20 | 40 | 9 | 7 | 18 | 30 | 18 | 12 | 4 | 4 | 12
Participants | 7 | 7 | 2 | 1 | 1 | 1 | 2 | 0 | 1 | 2 | 1 | 1 | 2

2. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MB-102
Description: Blood samples were collected pre-dose (time 0) and at 5, 10, 15; (± 1 or 2 min), 30, 60, 90, 120, 180, 240, 300 (±5 min), 360, 480, 600 and 720 (±10 min) minutes post dose, and were analyzed using validated analytical methods. Maximum plasma concentration (Cmax; measured in ng/mL) was directly determined from the concentration-time data.
Time Frame: Pre-dose and 5, 10, 15; (± 1 or 2 min), 30, 60, 90, 120, 180, 240, 300 (±5 min), 360, 480, 600 and 720 (±10 min) minutes post dose.
Population: All participants who received study drug and had no major protocol deviations.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) and 2 Doses MB-102: Two doses of MB-102 administered to participants 12 hours apart, with normal to chronic kidney disease (CKD) Stage 2 renal function, and fluorescence measured by the Brilliance ORFM device (1-2 sensors and 2-part sensor).The optimized algorithm and final device design of the Brilliance device was tested. Approximately half of the participants were to be enrolled with Fitzpatrick Scale Type I, II or III, and half with Type IV, V and VI skin color type.
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance | Normal-CKD Stage 2/Brilliance Algorithm Optimization | CKD Stage 3-5/Brilliance Algorithm Optimization | Normal-CKD Stage 2/Brilliance Sensor Optimization | Normal-CKD Stage 2/Brilliance Sensor Validation | CKD Stage 3-5/Brilliance Sensor Validation | Normal-CKD Stage 2/Brilliance (1-2 Sensors) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) and 2 Doses MB-102 | CKD Stage 3-5/Brilliance 1-2 Sensors
Number analyzed (Participants) | 31 | 29 | 20 | 40 | 9 | 7 | 18 | 30 | 18 | 12 | 4 | 4 | 12
ng/mL | 10751.613 (2279.3699) | 11625.517 (2491.4304) | 11981.7 (2659.9568) | 12243.45 (2563.5734) | 13961.111 (3326.5064) | 14440.143 (3049.767) | 13747.739 (2985.4673) | 13453.74 (3886.9335) | 13039.944 (3819.8448) | 13015.833 (2314.2462) | 15650 (4023.6799) | 13125 (2818.2441) | 11665 (3637.8803)

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Iohexol
Description: as for outcome 2
Time Frame: as for outcome 2
Population: All participants who received study drug and had no major protocol deviations. Per protocol, those in the Brilliance device group did not receive iohexol.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance
Number analyzed (Participants) | 31 | 29 | 20 | 40
ng/mL | 295967.742 (71088.9039) | 290172.414 (74285.6788) | 333000 (70799.9405) | 329200 (98658.229)

4. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of MB-102
Description: Blood samples were collected pre-dose (time 0) and at 5, 10, 15; (± 1 or 2 min), 30, 60, 90, 120, 180, 240, 300 (±5 min), 360, 480, 600 and 720 (±10 min) minutes post dose, and were analyzed using validated analytical methods. The time to maximum plasma concentration (Tmax; measured in minutes) was directly determined from the concentration-time data.
Time Frame: as for outcome 2
Population: All participants who received study drug and had no major protocol deviations.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance | Normal-CKD Stage 2/Brilliance Algorithm Optimization | CKD Stage 3-5/Brilliance Algorithm Optimization | Normal-CKD Stage 2/Brilliance Sensor Optimization | Normal-CKD Stage 2/Brilliance Sensor Validation | CKD Stage 3-5/Brilliance Sensor Validation | Normal-CKD Stage 2/Brilliance (1-2 Sensors) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) and 2 Doses MB-102 | CKD Stage 3-5/Brilliance 1-2 Sensors
Number analyzed (Participants) | 31 | 29 | 20 | 40 | 9 | 7 | 18 | 30 | 18 | 12 | 4 | 4 | 12
minutes | 7.258 (5.2976) | 5.862 (2.341) | 5.25 (1.118) | 5.875 (2.2325) | 5 (0) | 6.429 (2.4398) | 6.111 (2.7416) | 5.167 (0.9129) | 12.222 (27.0197) | 5 (0) | 5 (0) | 5 (0) | 25 (67.7227)

5. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Iohexol
Description: as for outcome 4
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance
Number analyzed (Participants) | 31 | 29 | 20 | 40
minutes | 9.194 (5.338) | 7.069 (3.1388) | 6.5 (2.3508) | 6.875 (2.7003)

6. Secondary Outcome: The Elimination Half-life of MB-102
Description: Blood samples were collected pre-dose (time 0) and at 5, 10, 15; (± 1 or 2 min), 30, 60, 90, 120, 180, 240, 300 (±5 min), 360, 480, 600 and 720 (±10 min) minutes post dose, and were analyzed using validated analytical methods. The elimination half-life (the time required for the concentration of the drug to reach half of its original value) was calculated as t1/2 λz= ln(2)/ λz.
Time Frame: as for outcome 2
Population: All participants who received study drug and had no major protocol deviations.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance | Normal-CKD Stage 2/Brilliance Algorithm Optimization | CKD Stage 3-5/Brilliance Algorithm Optimization | Normal-CKD Stage 2/Brilliance Sensor Optimization | Normal-CKD Stage 2/Brilliance Sensor Validation | CKD Stage 3-5/Brilliance Sensor Validation | Normal-CKD Stage 2/Brilliance (1-2 Sensors) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) and 2 Doses MB-102 | CKD Stage 3-5/Brilliance 1-2 Sensors
Number analyzed (Participants) | 31 | 29 | 20 | 40 | 9 | 7 | 18 | 30 | 18 | 12 | 4 | 4 | 12
minutes | 130.712 (33.5894) | 314.267 (151.5375) | 135.821 (26.0772) | 301.21 (183.0147) | 123.681 (25.4325) | 245.7 (51.3774) | 140.176 (22.2139) | 122.86 (14.6245) | 305.944 (105.6855) | 126.049 (20.65) | 147.117 (23.779) | 127.842 (22.9881) | 440.488 (294.5741)

7. Secondary Outcome: The Elimination Half-life of Iohexol
Description: as for outcome 6
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance
Number analyzed (Participants) | 31 | 29 | 20 | 40
minutes | 148.056 (38.2236) | 366.529 (191.4136) | 151.776 (31.4044) | 347.574 (214.8895)

8. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration for MB-102
Description: Blood samples were collected pre-dose (time 0) and at 5, 10, 15; (± 1 or 2 min), 30, 60, 90, 120, 180, 240, 300 (±5 min), 360, 480, 600 and 720 (±10 min) minutes post dose, and were analyzed using validated analytical methods. The area under the plasma concentration-time curve (ng*min/mL) was be estimated from time 0 to the last measurable concentration using noncompartmental analyses.
Time Frame: as for outcome 2
Population: All participants who received study drug and had no major protocol deviations.
Measure: Mean (Standard Deviation); unit: ng*min/mL
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance | Normal-CKD Stage 2/Brilliance Algorithm Optimization | CKD Stage 3-5/Brilliance Algorithm Optimization | Normal-CKD Stage 2/Brilliance Sensor Optimization | Normal-CKD Stage 2/Brilliance Sensor Validation | CKD Stage 3-5/Brilliance Sensor Validation | Normal-CKD Stage 2/Brilliance (1-2 Sensors) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) and 2 Doses MB-102 | CKD Stage 3-5/Brilliance 1-2 Sensors
Number analyzed (Participants) | 31 | 29 | 20 | 40 | 9 | 7 | 18 | 30 | 18 | 12 | 4 | 4 | 12
ng*min/mL | 1131336.448 (254801.4255) | 2419911.379 (708114.7104) | 1211931.882 (296491.1469) | 2467846.174 (843410.9665) | 1121973.694 (190118.8591) | 2560133.925 (519858.5738) | 1235178.035 (310587.5336) | 1072786.062 (281421.3481) | 2476458.456 (543445.259) | 1384887.303 (345784.1469) | 1488269.994 (108723.6082) | 1316506.556 (314196.0436) | 3678411.381 (1344727.8138)

9. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration for Iohexol
Description: as for outcome 8
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*min/mL
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance
Number analyzed (Participants) | 31 | 29 | 20 | 40
ng*min/mL | 33329159.548 (7909842.8639) | 58097567.569 (15177720.419) | 36677146.278 (10789963.956) | 70005450.758 (30243153.821)

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity for MB-102
Description: Blood samples were collected pre-dose (time 0) and at 5, 10, 15; (± 1 or 2 min), 30, 60, 90, 120, 180, 240, 300 (±5 min), 360, 480, 600 and 720 (±10 min) minutes post dose, and were analyzed using validated analytical methods. The area under the plasma concentration-time curve (ng*min/mL) from time 0 to infinity was calculated as: AUC∞ = AUClast + LQC/λz where LQC is the predicted concentration (based on the terminal regression) at the time of the last measurable concentration.
Time Frame: as for outcome 2
Population: All participants who received study drug and had no major protocol deviations.
Measure: Mean (Standard Deviation); unit: ng*min/mL
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance | Normal-CKD Stage 2/Brilliance Algorithm Optimization | CKD Stage 3-5/Brilliance Algorithm Optimization | Normal-CKD Stage 2/Brilliance Sensor Optimization | Normal-CKD Stage 2/Brilliance Sensor Validation | CKD Stage 3-5/Brilliance Sensor Validation | Normal-CKD Stage 2/Brilliance (1-2 Sensors) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) and 2 Doses MB-102 | CKD Stage 3-5/Brilliance 1-2 Sensors
Number analyzed (Participants) | 31 | 29 | 20 | 40 | 9 | 7 | 18 | 30 | 18 | 12 | 4 | 4 | 12
ng*min/mL | 1166655.776 (298807.3587) | 3212036.698 (1490329.1808) | 1242760.175 (321230.0672) | 3045719.769 (1625406.4454) | 1182254.364 (208571.1669) | 2914852.088 (684490.5106) | 1264462.94 (333601.038) | 1086390.141 (287588.9895) | 3135394.594 (1051071.597) | 1403855.606 (355269.4445) | 1518516.431 (106177.2201) | 1340051.2 (332392.6494) | 3844963.027 (1630799.1909)

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity for Iohexol
Description: as for outcome 10
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*min/mL
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance
Number analyzed (Participants) | 31 | 29 | 20 | 40
ng*min/mL | 34688858.452 (9029243.5529) | 81061044.851 (37977572.641) | 38032869.839 (11788838.136) | 90107803.206 (61220389.979)

12. Secondary Outcome: Total Plasma Clearance of MB-102
Description: Blood samples were collected pre-dose (time 0) and at 5, 10, 15; (± 1 or 2 min), 30, 60, 90, 120, 180, 240, 300 (±5 min), 360, 480, 600 and 720 (±10 min) minutes post dose, and were analyzed using validated analytical methods. Total plasma clearance (the volume of plasma cleared of the drug over time) was calculated as: Clp = Dose/ AUC∞.
Time Frame: as for outcome 2
Population: All participants who received study drug and had no major protocol deviations.
Measure: Mean (Standard Deviation); unit: mL/minute
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance | Normal-CKD Stage 2/Brilliance Algorithm Optimization | CKD Stage 3-5/Brilliance Algorithm Optimization | Normal-CKD Stage 2/Brilliance Sensor Optimization | Normal-CKD Stage 2/Brilliance Sensor Validation | CKD Stage 3-5/Brilliance Sensor Validation | Normal-CKD Stage 2/Brilliance (1-2 Sensors) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) and 2 Doses MB-102 | CKD Stage 3-5/Brilliance 1-2 Sensors
Number analyzed (Participants) | 31 | 29 | 20 | 40 | 9 | 7 | 18 | 30 | 18 | 12 | 4 | 4 | 12
mL/minute | 110.719 (28.2476) | 51.741 (21.4424) | 102.361 (31.8835) | 51.322 (26.2932) | 103.107 (17.1532) | 44.677 (13.798) | 97.496 (18.6913) | 117.913 (39.4472) | 42.838 (13.1284) | 99.216 (33.0196) | 84.29 (5.0376) | 97.741 (23.5163) | 38.736 (13.87)

13. Secondary Outcome: Total Plasma Clearance of Iohexol
Description: as for outcome 12
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/minute
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance
Number analyzed (Participants) | 31 | 29 | 20 | 40
mL/minute | 97.596 (22.6026) | 47.418 (19.9867) | 90.788 (25.7641) | 45.963 (19.1755)

14. Secondary Outcome: The Terminal Rate Constant for MB-102
Description: Blood samples were collected pre-dose (time 0) and at 5, 10, 15; (± 1 or 2 min), 30, 60, 90, 120, 180, 240, 300 (±5 min), 360, 480, 600 and 720 (±10 min) minutes post dose, and were analyzed using validated analytical methods. The terminal rate constant (λz) was determined by linear regression of the terminal linear phase of the log plasma concentration-time profile.
Time Frame: as for outcome 2
Population: All participants who received study drug and had no major protocol deviations.
Measure: Mean (Standard Deviation); unit: 1/minutes
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance | Normal-CKD Stage 2/Brilliance Algorithm Optimization | CKD Stage 3-5/Brilliance Algorithm Optimization | Normal-CKD Stage 2/Brilliance Sensor Optimization | Normal-CKD Stage 2/Brilliance Sensor Validation | CKD Stage 3-5/Brilliance Sensor Validation | Normal-CKD Stage 2/Brilliance (1-2 Sensors) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) and 2 Doses MB-102 | CKD Stage 3-5/Brilliance 1-2 Sensors
Number analyzed (Participants) | 31 | 29 | 20 | 40 | 9 | 7 | 18 | 30 | 18 | 12 | 4 | 4 | 12
1/minutes | 0.006 (0.0012) | 0.003 (0.001) | 0.005 (0.0009) | 0.003 (0.0012) | 0.006 (0.001) | 0.003 (0.0007) | 0.005 (0.0008) | 0.006 (0.0006) | 0.003 (0.0009) | 0.006 (0.0009) | 0.005 (0.0008) | 0.006 (0.0009) | 0.002 (0.0007)

15. Secondary Outcome: The Terminal Rate Constant for Iohexol
Description: as for outcome 14
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 1/minutes
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance
Number analyzed (Participants) | 31 | 29 | 20 | 40
1/minutes | 0.005 (0.001) | 0.002 (0.0009) | 0.005 (0.0009) | 0.002 (0.0008)

16. Secondary Outcome: Renal Clearance of MB-102
Description: Urine samples were collected pre-dose (time 0) and 5 mL urine samples were collected each time the subject voided. The total volume of urine excreted was recorded until 12 hours post-dose, and was analyzed using validated analytical methods. Renal clearance (the volume of plasma cleared of the drug by the kidneys over time) was calculated as: CLr = Ae/ AUClast, where Ae is the cumulative amount of analyte excreted in urine over the sampling interval.
Time Frame: Pre-dose and each time the participant voids up to 720 minutes post dose
Population: All participants who received study drug and had no major protocol deviations.
Measure: Mean (Standard Deviation); unit: mL/minute
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance | Normal-CKD Stage 2/Brilliance Algorithm Optimization | CKD Stage 3-5/Brilliance Algorithm Optimization | Normal-CKD Stage 2/Brilliance Sensor Optimization | Normal-CKD Stage 2/Brilliance Sensor Validation | CKD Stage 3-5/Brilliance Sensor Validation | Normal-CKD Stage 2/Brilliance (1-2 Sensors) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) and 2 Doses MB-102 | CKD Stage 3-5/Brilliance 1-2 Sensors
Number analyzed (Participants) | 31 | 29 | 20 | 40 | 9 | 7 | 18 | 30 | 17 | 12 | 4 | 4 | 12
mL/minute | 111.396 (27.9973) | 52.171 (21.825) | 104.008 (32.3622) | 51.915 (26.3905) | 105.144 (19.2031) | 45.397 (14.1766) | 99.072 (19.0079) | 120.452 (40.0937) | 42.51 (12.9745) | 109.924 (35.5733) | 88.795 (3.2184) | 103.774 (24.9108) | 38.373 (13.0747)

17. Secondary Outcome: Renal Clearance of Iohexol
Description: as for outcome 16
Time Frame: Pre-dose and each time the participant voids up to 720 minutes post dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/minute
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance
Number analyzed (Participants) | 31 | 29 | 20 | 40
mL/minute | 98.548 (22.5239) | 47.909 (20.1816) | 92.258 (26.5401) | 46.109 (19.4391)

18. Secondary Outcome: Correlation Between the Transdermal Fluorescence Intensity of MB-102 as Measured by the Quantum Leap Device and Plasma Concentration of MB-102 at Each Time Point in the Renal Excretion Phase
Description: Blood samples were collected pre-dose (time 0) and at 5, 10, 15; (± 1 or 2 min), 30, 60, 90, 120, 180, 240, 300 (±5 min), 360, 480, 600 and 720 (±10 min) minutes post dose, and were analyzed using validated analytical methods. Transdermal fluorescence intensity at the time of blood sampling as measured by the QuantumLeap device was documented, and the correlation between the transdermal fluorescence intensity of MB-102 as measured by the QuantumLeap device and the plasma concentration of MB-102 at each time point in the renal excretion phase was calculated.
Time Frame: Pre-dose (time 0) and 5, 10, 15; (± 1 or 2 min), 30, 60, 90, 120, 180, 240, 300 (±5 min), 360, 480, 600 and 720 (±10 min) minutes post dose
Population: All participants who received study drug and had no major protocol deviations
Measure: Mean (Standard Deviation); unit: Coefficient of determination, r-squared
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap
Number analyzed (Participants) | 31 | 29
Coefficient of determination, r-squared | -0.999 (0.0009) | -0.998 (0.0028)

19. Secondary Outcome: Correlation Between the Transdermal Fluorescence Intensity of MB-102 as Measured by the Radiance Device and Plasma Concentration of MB-102 at Each Time Point in the Renal Excretion Phase
Description: Blood samples were collected pre-dose (time 0) and at 5, 10, 15; (± 1 or 2 min), 30, 60, 90, 120, 180, 240, 300 (±5 min), 360, 480, 600 and 720 (±10 min) minutes post dose, and will be analyzed using validated analytical methods. Transdermal fluorescence intensity at the time of blood sampling as measured by the Radiance device was documented, and the correlation between the transdermal fluorescence intensity of MB-102 as measured by the Radiance device and the plasma concentration of MB-102 at each time point in the renal excretion phase was calculated.
Time Frame: as for outcome 18
Population: All participants who received study drug and had no major protocol deviations
Measure: Mean (Standard Deviation); unit: Coefficient of determination, r-squared
Arm/Group | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance
Number analyzed (Participants) | 20 | 40
Coefficient of determination, r-squared | -0.999 (0.001) | -0.998 (0.0033)

20. Secondary Outcome: Correlation Between the Transdermal Fluorescence Intensity of MB-102 as Measured by the Brilliance Device and Plasma Concentration of MB-102 at Each Time Point in the Renal Excretion Phase in Participants With Normal-CKD Stage 2 Renal Function
Description: Blood samples were collected pre-dose (time 0) and at 5, 10, 15; (± 1 or 2 min), 30, 60, 90, 120, 180, 240, 300 (±5 min), 360, and 480 minutes post dose, and were analyzed using validated analytical methods. Transdermal fluorescence intensity at the time of blood sampling as measured by the Brilliance device was documented, and the correlation between the transdermal fluorescence intensity of MB-102 as measured by the Brilliance device and the plasma concentration of MB-102 at each time point in the renal excretion phase was calculated.
Time Frame: Pre-dose (time 0) and 5, 10, 15; (± 1 or 2 min), 30, 60, 90, 120, 180, 240, 300 (±5 min), 360, and 480 minutes post dose
Population: All participants who received study drug and had no major protocol deviations
Measure: Mean (Standard Deviation); unit: Coefficient of determination, r-squared
Arm/Group | Normal-CKD Stage 2/Brilliance Algorithm Optimization | Normal-CKD Stage 2/Brilliance Sensor Optimization | Normal-CKD Stage 2/Brilliance Sensor Validation | Normal-CKD Stage 2/Brilliance (1-2 Sensors) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) and 2 Doses MB-102
Number analyzed (Participants) | 9 | 18 | 30 | 12 | 4 | 4
Coefficient of determination, r-squared | -0.994 (0.0092) | -0.998 (0.0026) | -0.999 (0.0015) | -0.997 (0.0037) | -0.999 (0.0015) | -1 (0.0001)

21. Secondary Outcome: Correlation Between the Transdermal Fluorescence Intensity of MB-102 as Measured by the Brilliance Device and Plasma Concentration of MB-102 at Each Time Point in the Renal Excretion Phase in Participants With CKD Stage 3-4 Renal Function
Description: Blood samples were collected pre-dose (time 0) and at 5, 10, 15; (± 1 or 2 min), 30, 60, 90, 120, 180, 240, 300 (±5 min), 360, 480, 600 and 720 (±10 min) and 960, 1440, 1920, 2400, and 2880 (±30 min) minutes post dose, and were analyzed using validated analytical methods. Transdermal fluorescence intensity at the time of blood sampling as measured by the Brilliance device was documented, and the correlation between the transdermal fluorescence intensity of MB-102 as measured by the Brilliance device and the plasma concentration of MB-102 at each time point in the renal excretion phase was calculated.
Time Frame: Pre-dose (time 0) and 5, 10, 15; (± 1 or 2 min), 30, 60, 90, 120, 180, 240, 300 (±5 min), 360, 480, 600 and 720 (±10 min) and 960, 1440, 1920, 2400, and 2880 (±30 min) minutes post dose
Population: All participants who received study drug and had no major protocol deviations
Measure: Mean (Standard Deviation); unit: Coefficient of determination, r-squared
Arm/Group | CKD Stage 3-5/Brilliance Algorithm Optimization | CKD Stage 3-5/Brilliance Sensor Validation | CKD Stage 3-5/Brilliance 1-2 Sensors
Number analyzed (Participants) | 7 | 18 | 12
Coefficient of determination, r-squared | -0.999 (0.0015) | -0.998 (0.0018) | -0.993 (0.0193)

22. Secondary Outcome: Number of Participants With Adverse Events Related to the Use of the QuantumLeap Device
Description: The number of participants with adverse events related to the use of the QuantumLeap device was documented.
Time Frame: From the time of dosing through the follow-up visit, up to 10 days
Population: Safety Analysis Set: all participants who signed the informed consent form and received study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap
Number analyzed (Participants) | 31 | 29
Participants | 4 | 0

23. Secondary Outcome: Number of Participants With Adverse Events Related to the Use of the Radiance Device
Description: The number of participants with adverse events related to the use of the Radiance device was documented.
Time Frame: From the time of dosing through the follow-up visit, up to 10 days
Population: Safety Analysis Set: all participants who signed the informed consent form and received study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance
Number analyzed (Participants) | 20 | 40
Participants | 1 | 0

24. Secondary Outcome: Number of Participants With Adverse Events Related to the Use of the Brilliance Device
Description: The number of participants with adverse events related to the use of the Brilliance device was documented.
Time Frame: From the time of dosing through the follow-up visit, up to 10 days
Population: Safety Analysis Set: all participants who signed the informed consent form and received study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Normal-CKD Stage 2/Brilliance Algorithm Optimization | CKD Stage 3-5/Brilliance Algorithm Optimization | Normal-CKD Stage 2/Brilliance Sensor Optimization | Normal-CKD Stage 2/Brilliance Sensor Validation | CKD Stage 3-5/Brilliance Sensor Validation | Normal-CKD Stage 2/Brilliance (1-2 Sensors) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) and 2 Doses MB-102 | CKD Stage 3-5/Brilliance 1-2 Sensors
Number analyzed (Participants) | 9 | 7 | 18 | 30 | 18 | 12 | 4 | 4 | 12
Participants | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the time of dosing through the follow-up visit, up to 10 days
Arm/Group | Normal-CKD Stage 2/QuantumLeap | CKD Stage 3-4/QuantumLeap | Normal-CKD Stage 2/Radiance | CKD Stage 3-5/Radiance | Normal-CKD Stage 2/Brilliance Algorithm Optimization | CKD Stage 3-5/Brilliance Algorithm Optimization | Normal-CKD Stage 2/Brilliance Sensor Optimization | Normal-CKD Stage 2/Brilliance Sensor Validation | CKD Stage 3-5/Brilliance Sensor Validation | Normal-CKD Stage 2/Brilliance (1-2 Sensors) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) and 2 Doses MB-102 | CKD Stage 3-5/Brilliance 1-2 Sensors
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29 | 0/20 | 0/40 | 0/9 | 0/7 | 0/18 | 0/30 | 0/18 | 0/12 | 0/4 | 0/4 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29 | 0/20 | 0/40 | 0/9 | 0/7 | 0/18 | 0/30 | 0/18 | 0/12 | 0/4 | 0/4 | 0/12
Other Adverse Events (participants affected / at risk) | 7/31 | 5/29 | 2/20 | 0/40 | 1/9 | 1/7 | 2/18 | 0/30 | 1/18 | 2/12 | 1/4 | 1/4 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal-CKD Stage 2/QuantumLeap (N=31) | CKD Stage 3-4/QuantumLeap (N=29) | Normal-CKD Stage 2/Radiance (N=20) | CKD Stage 3-5/Radiance (N=40) | Normal-CKD Stage 2/Brilliance Algorithm Optimization (N=9) | CKD Stage 3-5/Brilliance Algorithm Optimization (N=7) | Normal-CKD Stage 2/Brilliance Sensor Optimization (N=18) | Normal-CKD Stage 2/Brilliance Sensor Validation (N=30) | CKD Stage 3-5/Brilliance Sensor Validation (N=18) | Normal-CKD Stage 2/Brilliance (1-2 Sensors) (N=12) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) (N=4) | Normal-CKD Stage 2/Brilliance (1-2 Sensors and Brilliance 2-part Sensor) and 2 Doses MB-102 (N=4) | CKD Stage 3-5/Brilliance 1-2 Sensors (N=12)
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site discoloration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Application site erythema (General disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1
Oedema peripheral (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MediBeacon requests that no presentation/publication occur until after the first publication of study results or until 1 yr after a study is completed/terminated early, whichever occurs first. Proposed results publication/disclosure must be given to Sponsor for review at least 45 days prior to the date of submission. If a patent application is to be filed, both the Institution and the Sponsor will defer publication or other disclosure for a period of time, not to exceed an additional 60 days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT02772276/Prot_SAP_000.pdf